CLINICAL TRIAL: NCT06510491
Title: A Phase 2 Trial Investigating Epcoritamab in Patients With Previously Treated Waldenstrom Macroglobulinemia (WM)
Brief Title: Epcoritamab in Previously Treated WM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gottfried von Keudell, MD PhD (Other)
Collaborators: Genmab (Industry)
Responsible Party: Sponsor-Investigator, Gottfried von Keudell, MD PhD, Sponsor Investigator, Beth Israel Deaconess Medical Center
Organization: Beth Israel Deaconess Medical Center (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24-121
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Waldenstrom Macroglobulinemia; B-Cell Lymphoproliferative Disorder
Keywords: Waldenstrom Macroglobulinemia; B-Cell Lymphoproliferative Disorder
MeSH Terms: conditions — Waldenstrom Macroglobulinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Safety Lead-In Epcoritamab (Experimental): Participants will be enrolled using a modified 3+3 dose-escalation design to establish the Recommended Phase 2 Dose of Epcoritamab and will complete study procedures as follows:
  * Baseline visit with CT scan and bone marrow biopsy.
  * Bone marrow biopsy before cycle 6.
  * Cycles 1 - 3:
    --Days 1, 8, 15, and 22 of 28 day cycle: Predetermined dose of Epcoritamab 1x daily.
  * Cycles 4 - 9:
    --Days 1 and 15 of 28 day cycle: Predetermined dose of Epcoritamab 1x daily.
  * Cycles 10 - 12:
    --Day 1 of 28 day cycle: Predetermined dose of Epcoritamab 1x daily.
  * End of Treatment visit with CT scan and bone marrow biopsy.
  * Follow up visits: every 3 months for 2 years
  * Off study visit
  * If there are 0 out of 3 dose-limiting toxicities (DLTs), the study will proceed to phase II. If 1/3 participants experience a DLT, up to 3 additional participants will be treated at the same dose level. If more than 1/6 total participants experience a DLT, then the study will not proceed to phase 2.
  Interventions: Drug: Epcoritamab
- Phase II Epcoritamab (Experimental): Participants will be enrolled and will complete study procedures as follows:
  * Baseline visit with CT scan and bone marrow biopsy.
  * Bone marrow biopsy before cycle 6.
  * Cycles 1 - 3:
    --Days 1, 8, 15, and 22 of 28 day cycle: Predetermined dose of Epcoritamab 1x daily.
  * Cycles 4 - 9:
    --Days 1 and 15 of 28 day cycle: Predetermined dose of Epcoritamab 1x daily.
  * Cycles 10 - 12:
    --Day 1 of 28 day cycle: Predetermined dose of Epcoritamab 1x daily.
  * End of Treatment visit with CT scan and bone marrow biopsy.
  * Follow up visits: every 3 months for 2 years
  * Off study visit
  Interventions: Drug: Epcoritamab

INTERVENTIONS:
Drug: Epcoritamab — Bispecific antibody, via subcutaneous (under the skin) injection per protocol.
  Other Names: GEN3013; DuoBody-CD3xCD20

SUMMARY:
This study is being done to determine if epcoritamab can be used to treat participants with previously treated Waldenstrom Macroglobulinemia (WM).

The names of the study drug involved in this study is:

-Epcoritamab (a type of antibody)

DETAILED DESCRIPTION:
This is a prospective phase 2, single arm, open label trial to determine if epcoritamab can be used to treat participants with previously treated Waldenstrom Macroglobulinemia (WM). Epcoritamab is a bispecific antibody, a synthetic protein that activates the immune system to target cancer cells.

The U.S. Food and Drug Administration (FDA) has not approved epcoritamab for WM.

The research study procedures include screening for eligibility, in-clinic visits, questionnaires, blood tests, electrocardiograms, bone marrow biopsies, and Computerized Tomography (CT) scans.

Participants will receive study treatment for up to 4 months and will be followed for 24 months.

It is expected that about 20 people will take part in this research study.

Genmab, Inc. is funding this research study by providing the study drug, epcoritamab.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of lymphoplasmacytic lymphoma/WM that is CD20+ by immunophenotype or immunohistochemistry confirmed by bone marrow biopsy/aspirate (fresh or archival tissue acceptable) at time of most recent progression. All degrees of CD20 positivity will be accepted.
* Serum IgM level >2x upper limit of normal (ULN)
* Meeting criteria for initiation of treatment per IWWM2 criteria [Kyle Semin Oncol 2002], including but not limited to hyperviscosity syndrome, peripheral neuropathy, cold agglutinin disease, cryoglobulinemia, amyloidosis, cytopenias due to bone marrow infiltration, symptomatic or bulky lymph nodes, symptomatic splenomegaly, constitutional symptoms not otherwise explained by other causes, signs of organ dysfunction secondary to WM
* At least one prior line of treatment that was discontinued either due to intolerance or disease progression
* Prior therapies must have included an anti-CD20 antibody (e.g. rituximab) and a BTK inhibitor (e.g. ibrutinib, zanubrutinib). Patients who received ibrutinib and rituximab in combination as first line therapy will be eligible. BTKi should be stopped to allow a washout period of no less than 4 half-lives prior to epcoritamab.
* Age ≥18 years
* ECOG performance status £ 2
* Life expectancy of greater than 2 years
* Participants must meet the following organ and marrow function as defined below:

  * absolute neutrophil count ≥1000 cells/mcl (G-CSF allowed)
  * absolute lymphocyte count ≥200 cells/mcl
  * platelets ≥75,000 cells/mcl OR ≥50,000 cells/mcl in the presence of bone marrow involvement or splenomegaly (Note: no PLT transfusions within 7 days prior to screening)
  * hemoglobin ≥ 8 g/dL (transfusion allowed)
  * total bilirubin ≤ 1.5 institutional upper limit of normal (ULN). In patients with suspected/known Gilbert's disease total bilirubin up to 3x ULN will be allowed but direct bilirubin must be ≤ 2 x ULN
  * AST(SGOT)/ALT(SGPT) ≤3× institutional ULN
  * creatinine ≤ institutional ULN OR
  * creatinine clearance >45 ml/min (by Cockcroft-Gault estimate or 24-hr creatinine clearance measurement)
* Subject does not have an active (PCR-positive) Hepatitis B virus (HBV) or Hepatitis C virus (HCV) infection. If laboratory evidence for a chronic infection with hepatitis B, close monitoring and prophylactic therapy is required as described in Section 5.4.
* Participants with a history of prior malignancy will be eligible if all treatment of that malignancy was completed at least 2 years before registration, the treatment was considered "curable-intent", and there is no evidence of disease.
* Ability to understand and the willingness to sign a written informed consent document.
* Females of childbearing potential must agree to practice a highly effective method of birth control (as defined by the EU Clinical Trial Facilitation Group) consistent with local regulations regarding the use of birth control methods for patients participating in clinical trials:

  * Established use of oral, injected or implanted combined (estradiol and progesterone containing) hormonal contraception;
  * Placement of an intrauterine device (IUD) or intrauterine system (IUS);
  * Male partner sterilization (the vasectomized partner should be the sole partner for that patient)
  * True abstinence (when this is in line with the preferred and usual lifestyle of the patient)
* Women must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the trial and for 12 months after receiving the last dose of epcoritamab. Men must also not donate sperm during the trial and for 12 months after receiving the last dose of epcoritamab.
* A man who is sexually active with a woman of childbearing potential must agree to use a barrier method of birth control (i.e. use of condom) during the trial and for 12 months after receiving the last dose of epcoritamab.
* Patients with HIV may be enrolled if they are on stable antiretroviral therapy, have an undetectable viral load, and CD4 count > 250 cells/mm3.

Exclusion Criteria:

* Participants who have disease that has transformed to aggressive lymphoma
* Participants with symptomatic or suspected hyperviscosity syndrome or IgM levels greater than 4000 mg/dL who are unable to undergo plasmapheresis to decrease the risk of an IgM flare. Participants who can undergo plasmapheresis will be eligible as long as they undergo the procedure prior to first treatment dose.
* Participants who are receiving any other investigational agent
* Washout from prior therapy: BTKi: no less than5 half-lives prior to epcoritamab to prevent BTKi rebound and rituximab: no less than 4 weeks (28 days) from last dose.
* Participants who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) except for alopecia and peripheral neuropathy
* Uncontrolled intercurrent active infection requiring hospitalization or intravenous antimicrobial agents within 4 weeks of start of treatment
* Uncontrolled underlying cardiac conditions including but not limited to: congestive heart failure grade III or IV (by NYHA) or EF < 45%, unstable angina pectoris, acute myocardial infarction < 6 months, uncontrolled cardiac arrhythmia
* History of uncontrolled neurologic condition including but not limited to: seizure disorder, stroke, psychosis, dementia, CNS vasculitis, encephalitis
* Need for supplemental O2 at rest to maintain SaO2>92%
* Chronic immunosuppressive therapy for non-WM-related indication within 28 days of initiation of treatment, including systemic corticosteroids 20 mg/day or greater prednisone-equivalent
* Patients with known or suspected CNS involvement or leptomeningeal disease (i.e. BingNeel Syndrome) are excluded given concern for potentially increased risk of neurologic toxicity with epcoritamab. Patients with history of CNS malignancy from separate malignancy must have completed CNS-directed therapy and must currently have no evidence of disease
* Pregnant or breastfeeding women or participants unwilling to adhere to institutional guidelines for highly effective contraception for the duration of the therapy are excluded. This is because of the unknown but potential risk of teratogenic or abortifacient effects, as well as potential for adverse events in nursing infants secondary to treatment of the mother, as epcoritamab has not yet been studied in this patient population. A female can be determined to not be of childbearing potential if she meets any of the following criteria:

  * Premenarchal
  * Postmenopausal (>45 years of age with amenorrhea for at least 12 months or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone [FSH] level >40 IU/L or mIU/mL)
  * Permanently sterilized (e.g., bilateral tubal occlusion [which includes tubal ligation procedures as consistent with local regulations], hysterectomy, bilateral salpingectomy, bilateral oophorectomy) Note: If the childbearing potential changes after start of the trial (e.g., woman who is not heterosexually active becomes active, premenarchal woman experiences menarche) a woman must begin a highly effective method of birth control, as described under 3.1.13.
* Known current alcohol or drug abuse, psychiatric illness, or unstable social situation that is likely to limit compliance with study requirements
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to epcoritamab
* Exposure to a live or a live attenuated vaccine within 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to 12 cycles of treatment (28 days per cycle)
  The overall response rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) based on modified IWWM6 criteria.

SECONDARY OUTCOMES:
6-month Best Response Rate | 6 months
  Best response on treatment was based on modified IWWM6 criteria. Including complete response (CR), very good partial response (VGPR), partial response (PR), stable disease (SD) and progressive disease (PD). Rate defined as the proportion of participants achieving the certain response.
Major Response Rate (MRR) | Up to 12 cycles of treatment (28 days per cycle)
  MMR defined as proportion pf participants achieving the major response includes PR, VGPR, and CR based on IWWM6 criteria.
Median Time to Best Response | Up to 12 cycles of treatment (28 days per cycle)
  Best response on treatment was based on modified IWWM6 criteria. Time to event outcome estimate using Kaplan-Meier method.
Median Duration of Overall Response (DOR) | Up to 12 cycles of treatment (28 days per cycle)
  Duration of Overall Response (DOR), estimated using the Kaplan Meier method, is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) per modified IWWM6 criteria, until the first date that recurrent or progressive disease is objectively documented. Participants without progressive disease are censored at the date of last disease assessment.
2-year Progression-Free Survival (PFS) Rate | 2 years
  2-year PFS is a probability estimated using progression-free survival based on the Kaplan-Meier method is defined as the duration between registration and documented disease progression (PD) or death, or is censored at time of last disease assessment.
Median Time to Next Line of Therapy (TTNT) | Up to 2 years
  Kaplan-Meir method will be used to estimate the TTNT. TTNT is defined as period of time from initiation of epcoritamab until start of next line of treatment.
2-year Overall Survival (OS) | 2 years
  2-year OS is a probability estimated using the Kaplan-Meier method; OS is defined as the time from study entry to death, or censored at date last known alive.
Grade 3-5 Treatment-related Toxicity Rate | Up to 12 cycles of treatment (28 days per cycle)
  All grade 3-5 adverse events (AE) with treatment attribution of possibly, probably or definite based on IWWM6 criteria that are not resolved in accordance with treatment guidelines were counted. Rate is the proportion of treated participants experiencing at least one of these adverse events as defined during the time of observation.

CONTACTS AND LOCATIONS:
Overall Officials: Gottfried von Keudell, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu